CLINICAL TRIAL: NCT01792206
Title: EFFECT OF PARICALCITOL (ZEMPLAR) ON ENDOTHELIAL FUNCTION AND INFLAMMATION IN TYPE 2 DIABETES AND CHRONIC KIDNEY DISEASE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Scott and White Hospital & Clinic (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Vasudevan Raghavan, Director, CArdioMEtabolic, Lipid Clinic and Medical Weight Management Program Services, Scott and White Hospital & Clinic
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 81890
Record Dates: First submitted 2012-02-29; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Type 2 Diabetes; Chronic Kidney Disease
Keywords: Stage 3 chronic kidney disease (CKD); Stage 4 chronic kidney disease (CKD); CKD
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic | interventions — paricalcitol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zemplar (Active Comparator): Zemplar 1 mcg or placebo to be taken once daily with breakfast for 3 months
  Interventions: Drug: Zemplar
- Placebo (Placebo Comparator): Zemplar 1 mcg or placebo to be taken once daily with breakfast for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zemplar — Zemplar 1 mcg or placebo to be taken once daily with breakfast for 3 months
  Arms: Zemplar
Drug: Placebo — Zemplar 1 mcg or placebo to be taken once daily with breakfast for 3 months
  Arms: Placebo

SUMMARY:
The purpose of this research study is to study the effects of paricalcitol on endothelial function and inflammation, cardiovascular risk factors which are associated with patient populations that have Type 2 diabetes and Stage 3 and 4 Chronic Kidney Disease (CKD).

Hypothesis 1: The state of CKD is associated with oxidative stress and inflammation and impaired post ischemic endothelium dependent flow mediated vasodilation which may contribute to atherogenesis.

Hypothesis 2: The administration of paracalcitol to patients with CKD will suppress oxidative stress and inflammation and improve endothelial function and thus contribute to an anti-atherogenic action.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Type 2 diabetes and CKD
2. Age 18 - 70 years
3. Stable anti-hypertensive and lipid lowering therapy for at least 2 months. All patients should be on an ACEI or ARB unless contraindicated because of side effects (standard of care). No changes in lipid lowering therapy during the 3 months of this study. Blood pressure doses may be changed but new therapy with ACE inhibitors will not be allowed.

Exclusion Criteria:

1. Severe co morbid conditions - e.g. Cancer, etc.
2. Congestive heart failure.
3. Inability to give informed consent or attend study related visits.
4. Have a history of abnormally high vitamin D or calcium levels in the bloodstream.
5. Unwilling or unable to complete screening or data collection procedures.
6. Have a known allergy to the study drug.
7. Pregnant or breast feeding
8. Plasma Calcium >9 mg/dl
9. Patients should discontinue any calcium supplementation prior to entry into the study.
10. Other vitamin D analogs (eg Sensipar) and vitamin D preparations are contraindicated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
The change in brachial artery Flow Mediated Dilataion with paracalcitol (1mcg/day)compared with placebo for 3 months. | Baseline, 4 weeks, and 12 weeks
  We therefore propose a study of the effects of Zemplar compared to placebo in patients with diabetes and stage 3-4 CKD on endothelial function and markers of inflammation and oxidative stress. The finding will help not only guide and encourage such treatment in similar patients, but will give us fundamental mechanistic insights into the role of vitamin D in the pathogenesis of diabetes and CVD.

SECONDARY OUTCOMES:
Biomarker Measurement | Baseline, 4 weeks, and 12 weeks
  Determine the prevalance of abnormalities in biomarkers of inflammation, oxidative stress and endothelial function in patients with CKD compared to a healthy population
  The following are the biomarkers of inflammation and oxidative stress to be measured in the secondary outcomes are:
  NFkB binding by mononuclear cells (MNC) ; ROS generation and p47phox expression by MNC plasma concentration of MMP-9, MCP-1, ICAM-1, IL-6 , CRP, ADMA and nitrotyrosine.. urinary isoprostane and plasma Nitrotyrosine in patients with CKD.
Biomarker Measurement | Baseline, 4 weeks, and 12 weeks
  Compare the change in biomarkers of inflammation, oxidative stress and endothelial function with paracalcitol (1mcg/day) compared with placebo for 3 months in patients with CKD.
  The following are the biomarkers of inflammation and oxidative stress to be measured in the secondary outcomes are:
  NFkB binding by mononuclear cells (MNC) ; ROS generation and p47phox expression by MNC plasma concentration of MMP-9, MCP-1, ICAM-1, IL-6 , CRP, ADMA and nitrotyrosine.. urinary isoprostane and plasma Nitrotyrosine in patients with CKD.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Emory University, Atlanta, Georgia
  - Tulane University, New Orleans, Louisiana
  - Joslin Diabetes Clinic, Inc., Boston, Massachusetts
  - Omaha VA Medical Center, Omaha, Nebraska